CLINICAL TRIAL: NCT04125316
Title: Level of FeNO in Chinese Asthma Patients
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fanny W.S. Ko, Honorary Clinical Associate Professor, Chinese University of Hong Kong
Other Study IDs: FeNO_study_protocol V1
Record Dates: First submitted 2019-09-27; First posted 2019-10-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma: Asthma patients
  Interventions: Other: Observation, no intervention

INTERVENTIONS:
Other: Observation, no intervention — Observational study, no intervnetion
  Other Names: No intervention

SUMMARY:
This study aims to assess the level of FeNO in Chinese asthma patients with respect to the different levels of asthma control over 1 year.

DETAILED DESCRIPTION:
Introduction Measurement of fractional nitric oxide (NO) concentration in exhaled breath (FeNO) has been shown to be a non-invasive, quantitative biomarker related to airway inflammation. Although there is inadequate evidence to support the use of FENO to aid the diagnosis of asthma, recent studies demonstrate the usefulness of FENO in phenotyping and management of asthma. American Thoracic Society (ATS) Clinical Practice Guideline recommended the use of FeNO in the diagnosis of eosinophilic airway inflammation and in determining the likelihood of steroid responsiveness in individuals with chronic respiratory symptoms possibly due to airway inflammation. The guideline recommends in adults with FENO less than 25 parts per billion (ppb) indicates eosinophilic inflammation and responsiveness to corticosteroids are less likely, and greater than 50 ppb indicates eosinophilic inflammation and, in symptomatic patients, responsiveness to corticosteroids are likely.

However, a validation study of ATS guideline showed almost one-fourth of patients had intermediate FENO values (i.e. 25-50ppb), which may limit the clinical usefulness of the ATS FeNO cut-points. Furthermore, FENO values are affected by multiple factors. In a recent study that assessed the determinants of FENO in men and women without lung diseases using data from 25 centres across 11 European countries and Australia involving 3881 subjects, it was found that gender, smoking status, height, IgE sensitization would affect the FeNO level measured.

A prior study also showed the FeNO levels of healthy Chinese children and adult without significant lung diseases are higher than the Caucasian population. An earlier genotyping findings of nitric oxide synthase genes suggested that the frequencies of minor alleles associated with nitric oxide production were substantially lower in Chinese subjects. Therefore, ethnic-specific references must be considered when setting the cut-off values for assessing asthma status in different populations.

There are many studies on the cut-off of FeNO for making a diagnosis of asthma. There are, however, not much information on the level of FeNO in Chinese asthma patients with different levels of asthma control in a real-life setting and whether the ATS clinical practice guideline is applicable for Chinese asthma subjects given that the healthy subjects had a higher FeNO than the Caucasian population.

The aim of this study is to assess the level of FeNO in Chinese asthma patients with respect to the different levels of asthma control over a period of 1 year.

Method Subject recruitment This is an observational study in which FeNO was measured in Chinese adults asthma patients in Hong Kong. Subjects will be recruited from the general medical and respiratory clinic of the Prince of Wales Hospital in Hong Kong. After an explanation of the study, the investigator will obtain the written informed consent from all the patients who meet the inclusion criteria and with no exclusion criteria.

Inclusion criteria:

• Chinese subjects aged between 18 and 90 years and have a diagnosis of asthma according to The Global Initiative for Asthma (GINA) guideline 2019. Asthma is defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 200 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable.

Exclusion criteria:

* Patients with respiratory diseases with other known respiratory diseases including chronic obstructive pulmonary disease, bronchiectasis, tuberculosis (TB)-destroyed lung parenchyma, history of lung resection and lung cancer
* Individuals older than 40 years with a smoking history of more than 10 pack-years
* Patients currently randomized in other clinical studies
* Pregnant women

In addition, healthy subjects with no respiratory symptoms and asthma as defined above, and other significant lung diseases, such as chronic obstructive pulmonary disease, history of tuberculosis and bronchiectasis) with normal CXR will be recruited as control subjects.

Assessment of the subjects:

After recruitment, asthma patient will be followed up in the research clinic every 4 months for one year. Patients will have the following assessment in each visit.

1. Demographic characteristics of the subjects Demographic characteristics of the subjects will include age, body weight and height, symptoms, age of onset of disease, exacerbations or hospital admission in the past 12 months for asthma, medications taking and vaccinations in the past 12 months.
2. FeNO measurement FeNO will be measured before spirometry. FeNO will be measured online using a NIOX VERO (Circassia, Oxford, UK) according to ATS/ERS recommendations. Subjects will be in the sitting position (with no nose clip), exhale to residual volume, insert a mouthpiece, inhale to total lung capacity, and then exhale for 10 seconds at a constant flow rate of 50mL/s. The measurement will be repeated until three FeNO values varied less than 10% or two values varied less than 5%. The mean FeNO (in ppb) will then be recorded. All subjects have to refrain from strenuous physical activity or exercise for at least 30 minutes prior to FeNO measurement. In addition, subjects shall avoid eating for 1 hour and caffeine ingestion for 6 hours before the test. Subjects will not be tested within 4 weeks of an upper or lower respiratory tract infection.
3. Spirometry pre- and post-bronchodilator Spirometry pre- and post-bronchodilator according to the American Thoracic Society and European Respiratory Society standards will be performed.14 The updated predicted spirometry values for Hong Kong Chinese will be used to calculate the predicted lung function.ong Kong Chinese will be used to calculate the predicted lung function.
4. Home peak expiratory flow rate (PEFR) monitoring Patients will be asked to measure their home PEFR using a PEFR monitoring meter (Mini-Wright, Clement Clarke International Ltd, Essex, UK) and will be asked to record their PEFR as the best of three recordings in the morning before the use of inhalers. Mean PEFR is the mean of the daily PEFR for the 2 weeks before the follow-up. PEFR variability was calculated using the Min%Max index (minimum PEFR, expressed as a percent of the best PEFR over 2 weeks before follow up).
5. Forced Oscillatory assessment of airway resistance Airway resistance and reactance will be assessed using the TremoFlo C-100 (Thrasys, Halifax, Canada). Forced oscillatory measures the resistance and reactance of the respiratory system during tidal breathing by superimposing a gentle multi-frequency airwave onto the patient's respiratory airflow. The parameters of airway resistance measured will include low-frequency resistance at 5 Hz denoted as R5 and difference from 5 Hz to 19 Hz denoted as R5 to R19. Low-frequency reactance at 5 Hz is denoted as X5, resonant frequency when elasticity balances inertia (i.e. Fres) and the low-frequency reactance area (i.e. ALX) are reactance parameters being assessed in the study.
6. Blood test Routine blood test, including blood eosinophil count and total IgE level as determined by clinical need.
7. Skin prick test Skin prick test was performed with a panel of allergen extracts including cat, dog, dermatophagoides pteronyssinus and D. farinae, Aspergillus, Mold Mix, Tree Mix and cockroach. A minimum wheal size of 3 mm will be defined as a positive response.
8. Assessment of asthma control Asthma control in the past 4 weeks will be assessed. They will be evaluated and classified into different levels of asthma symptom control, according to GINA 201914 (appendix 1). The asthmatic attacks that required courses of systemic steroid or hospitalization will be documented (by asking the patient and also checking with health records). In addition, Asthma Control Test and Asthma control questionnaire will be used to assess asthma control.

For control subject, they will attend the research clinic once to have assessments of demographic characteristics, FENO level, spirometry, airway resistance, blood and skin test as described above.

Primary endpoint of the study: FeNO level in Chinese asthma of different levels of asthma control.

Secondary endpoint: FeNO level and risk of exacerbation in the subsequent 12 months, correlation of FeNO with makers of atopy and lung function including skin prick test, IgE level, eosinophil level and lung function parameters (spirometry and airway resistance).

Statistics Data will be analyzed by the Statistical Package of the Social Science Statistical software (SPSS) for Window, Version 22.0.0 (IBM SPSS Inc, IL, USA). The clinical characteristics of the subjects will be expressed as mean (SD) for normally distributed parameters or median (IQR) for non-normally distributed ones. FeNO levels between different levels of asthma control will be assessed by one-way ANOVA, while within individual variations with regard to the level of control and over time will be assessed by ANOVA with repeated measures, adjusted by age, sex, height and presence of atopy. Comparison of the FeNO levels of the asthma and control group will be assessed by independent sample t-test. Levels of FENO and time to first exacerbation will be assessed by Cox proportional-hazards model and log-rank test as appropriate. A p-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Chinese subjects aged between 18 and 90 years, and
* Have a diagnosis of asthma according to The Global Initiative for Asthma (GINA) guideline 2019. Asthma is defined as those with a consistent history and prior documented evidence of variable airflow obstruction, with evidence of an increase in FEV1 greater than 12% or 200 mL following bronchodilator or bronchial hyperresponsiveness on bronchial provocation testing, when stable.

Exclusion Criteria:

* Patients with respiratory diseases with other known respiratory diseases including chronic obstructive pulmonary disease, bronchiectasis, tuberculosis (TB)-destroyed lung parenchyma, history of lung resection and lung cancer
* Individuals older than 40 years with a smoking history of more than 10 pack-years
* Patients currently randomized in other clinical studies
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients attending clinic at the Prince of Wales Hospital in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
the level of FeNO | 1 year
  to assess the level of FeNO in Chinese asthma patients with respect to the different levels of asthma control over a period of 1 year.

SECONDARY OUTCOMES:
FeNO and risk of asthma exacerbation | 1 year
  FeNO level in ppb and number of asthma exacerbation in the subsequent 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan